CLINICAL TRIAL: NCT04110795
Title: Personalizing Osteoporosis Care: Clinical & Genetic Risk Factors for Atypical Femur Fractures
Brief Title: Personalizing Osteoporosis Care: Clinical & Genetic Risk Factors for AFFs
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 18-6171
Record Dates: First submitted 2019-09-25; First posted 2019-10-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Atypical Femur Fracture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood samples serum samples fingernail samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Atypical Femur fracture cases
  Interventions: Other: No Intervention
- Control: matched to AFF cases by race, age, length of ART use
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The overall objective of this project is to identify clinical and genetic risk factors for Atypical Femur Fractures (AFFs) in Anti-resorptive therapy (ART) users by conducting a case control study of 330 cases of AFFs and 660 controls without AFFs matched for age, sex, race and duration of ART.

DETAILED DESCRIPTION:
Antiresorptive therapy (ART) drugs are effective osteoporosis treatment and help decrease osteoporosis-related fractures. However, their long-term use has been associated with rare but serious atypical femur fractures (AFFs). Fear of these side effects has caused a substantial decline in the use of these effective drugs and rising fracture rates. The investigators propose to compare 330 cases of people with AFFs to 660 matched controls to explore similarities and differences in (1) clinical findings, such as type of ART and length of use, prior fracture, bone density, femur geometry, etc., and (2) genetic variants, and then (3) to validate the top few genetic variants to see if they are indeed present in an additional group of 100 AFF patients and not present in 100 control subjects. This study will determine clinical and genetic risk factors for these debilitating atypical fractures such that at-risk patients in the future can be treated differently to avoid them.

ELIGIBILITY:
Inclusion Criteria:

* Cases: Have experienced a confirmed, documented Atypical femur fracture
* Controls: currently on anti-resorptive therapy, matches AFF case by age, race and length of ART use

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community based population in Ontario and British Columbia Canada
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Associations between AFF and clinical Risk Factor | baseline
  Associations between AFFs and clinical risk factors
Associations between AFF and common genetic variants | baseline
  Associations of common genetic variants among patients with AFFs
Validation of top genetic variants | baseline
  To validate the top few genetic variants identified in the above case-control study in a separate cohort of 100 cases and 100 controls.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Cheung, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - Adachi Medical Centre, Hamilton, Ontario
  - Bone Research & Education Centre, Oakville, Ontario
  - University Health Network, TGH, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided